CLINICAL TRIAL: NCT03087578
Title: Comparison of Electroacupuncture to Mirabegron on Symptoms of Overactive Bladder in Women Who Have Failed Anti-Cholinergic Therapy
Brief Title: Comparison of Electroacupuncture to Mirabegron for Treatment of Overactive Bladder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHClevelandMC
Record Dates: First submitted 2017-03-13; First posted 2017-03-22 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Overactive Bladder
Keywords: overactive bladder, acupuncture
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EA (Experimental): Patients undergoing electroacupuncture weekly for 6 weeks for 30 minutes/session.
  Interventions: Other: electroacupncture
- Medication (Active Comparator): Patients will receive 50 mg of mirabegron daily for 6 weeks. Patients may continue to take this medication after the study if they have improvement in symptoms.
  Interventions: Drug: Mirabegron 50 MG [Myrbetriq]

INTERVENTIONS:
Other: electroacupncture — Patients will receive electroacupuncture treatment for 30 minutes per weekly session for 6 weeks.
  Arms: EA
Drug: Mirabegron 50 MG [Myrbetriq] — Patients will receive 50 mg of mirabegron daily for 6 weeks.
  Arms: Medication

SUMMARY:
This study compares electroacupuncture to mirabegron for treatment of overactive bladder (OAB) symptoms in women who have failed treatment with anticholingeric therapy.

DETAILED DESCRIPTION:
Screening/Eligibility Visit:

If it is determined that a patient with a diagnosis of OAB has failed therapy with at least one anti-cholinergic agent, the potential participant will be screened and eligibility will be confirmed by a study investigator. A signed, IRB-approved informed consent will be obtained.

Randomization:

Randomization will be performed after the patient has agreed to participate and discussed and signed the informed consent form. Patients will be randomized in random blocks of 4, 6 and 8 into either the acupuncture group or mirabegron group. Once patient participation is confirmed, an enveloped marked with the study participant number will be opened by one of the study investigators in front of the patient.

Acupuncture Protocol:

All acupuncture sessions will be performed by a licensed acupuncturist employed by University Hospitals Connor Integrative Health Network. All acupuncturists involved in the study protocol will be trained and supervised in the correct technique by Christine Kaiser, MS, LAc, Dipl.OM. Acupuncture session will be performed weekly for 6 weeks and will be scheduled to accommodate both the patient's and acupuncturists' schedules. Acupuncture sessions will last for 30 minutes. Selected points will include kidney 3, kidney 6, spleen 6, and ren 4. The current delivery with electroacupuncture is approximately 10-20 mA (adjusted to patient sensation) delivery at 10 Hz for 30 minutes per session. After completion of 6 weeks of treatments patients will be contacted by phone at 2 week intervals to determine duration of symptomatic relief after cessation of treatment..

Mirabegron Protocol:

Patients assigned to the medication group will be prescribed 50 mg of myrbetriq daily to take for 6 weeks. At the completion of the study, if patients are satisfied with the effect of mirabegron they may continue to use it at their discretion.

ELIGIBILITY:
Inclusion Criteria:

* - Patients must be 18 years or older as well as willing and able to provide informed consent
* Patients with documented symptoms of overactive bladder including: urgency, frequency >7 times per day, nocturia, urgency incontinence for at least 6 months
* Patients who have failed at least one anti-cholinergic medication defined as no change or unsatisfactory improvement in symptom severity after 6 weeks of a daily regimen

Exclusion Criteria:

* Patients younger than 18 years,
* Patients unable or unwilling to provide informed consent,
* Patients who are illiterate,
* Patients who are non-English speaking or reading,
* Patients with a current urinary tract infection
* Patients with a history of interstitial cystitis
* Patients who have a history of a bleeding disorder
* Patients who are currently on chronic anti-coagulation
* Patients who are have taken mirabegron in the past or are currently using it
* Patients currently undergoing acupuncture treatment for a different condition
* Patients who are currently undergoing pelvic floor physical therapy
* Patients who are currently undergoing or will undergo treatment for a urologic or gynecologic malignancy
* Patients who are currently pregnant
* Patients with an implanted pacemaker or AICD
* Patients with a history of uncontrolled or poorly controlled hypertension

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Difference in Incontinence Impact Questionnaire (IIQ-7) scores | at baseline, 3 weeks after therapy initiation, 6 weeks after therapy initiation, and monthly intervals for 3 months from therapy initiation for the acupuncture group
  change in IIQ-7 scores before and after initiation of treatment
Difference in Overactive Bladder Symptom Score (OABSS) | at baseline, 3 weeks after therapy initiation, 6 weeks after therapy initiation, and monthly intervals for 3 months from therapy initiation for the acupuncture group
  change in OABSS before and after initiation of treatment
Urogenital Distress Inventory (UDI-6) scores | at baseline, 3 weeks after therapy initiation, 6 weeks after therapy initiation, and monthly intervals for 3 months from therapy initiation for the acupuncture group
  change in UDI-6 scores before and after initiation of treatment
Differences in daytime frequency | at baseline, 3 weeks after therapy initiation, 6 weeks after therapy initiation, and monthly intervals for 3 months from therapy initiation for the acupuncture group
  before and after treatment
incontinence episodes | at baseline, 3 weeks after therapy initiation, 6 weeks after therapy initiation, and monthly intervals for 3 months from therapy initiation for the acupuncture group
  change in number of incontinence episodes before and after treatment
Nocturia | at baseline, 3 weeks after therapy initiation, 6 weeks after therapy initiation, and monthly intervals for 3 months from therapy initiation for the acupuncture group
  change in number of nocturia episodes before and after treatment

SECONDARY OUTCOMES:
Recurrence/worsening of symptoms | at baseline, 3 weeks after therapy initiation, 6 weeks after therapy initiation, and monthly intervals for 3 months from therapy initiation for the acupuncture group
  Recurrence/worsening of symptoms after cessation of acupuncture treatment

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hargreaves E, Baker K, Barry G, Harding C, Zhang Y, Kandala NB, Zhang X, Kernohan A, Clarkson CE. Acupuncture for treating overactive bladder in adults. Cochrane Database Syst Rev. 2022 Sep 23;9(9):CD013519. doi: 10.1002/14651858.CD013519.pub2. PMID 36148895